CLINICAL TRIAL: NCT05028894
Title: 23andMe Idiopathic Pulmonary Fibrosis Research Study
Brief Title: 23andMe IPF Research Study
Acronym: IPF
Status: Completed | Type: Observational
Sponsor: 23andMe, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 23andMe_IPF001
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; IPF; pulmonary fibrosis; lung diseases; lung; respiratory tract diseases; rare; rare diseases; Hermansky-Pudlak syndrome; HPS
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases; Rare Diseases; Hermanski-Pudlak Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Saliva sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IPF: Participants diagnosed with idiopathic pulmonary fibrosis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The long term goal of this study is to increase genetic understanding of IPF to enable the development of an effective drug for IPF that can improve the lives of those living with the condition.

DETAILED DESCRIPTION:
This study will recruit 1,000 people who have been diagnosed with IPF or Hermansky-Pudlak syndrome (HPS). Eligible participants who consent to participate in 23andMe Research and the IPF Research Study will receive a 23andMe Health + Ancestry kit at no cost. Participants will provide a saliva sample and take a baseline survey online answering questions about their disease diagnosis, testing, treatment, and symptoms. Participants will also be asked to take the same survey 3, 6, and 9 months after completing the baseline survey. The data collected from this study will be incorporated into the 23andMe Database and used to better understand the underlying genetic and environmental factors that contribute to IPF.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with IPF or Hermansky-Pudlak syndrome (HPS)
* Are 18+ years old
* Live in the US

Exclusion Criteria:

- Have been diagnosed with sarcoidosis or hypersensitivity pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will only include participants who meet the eligibility criteria as described above. Participants in the study will be diagnosed with IPF or HPS.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
IPF Symptom Progression Baseline | Baseline
  Survey asking about disease diagnosis, testing, treatments, and symptom progression
IPF Symptom Progression 3 month follow-up | 3 months post baseline
  IPF Symptom Progression 3 month follow-up
IPF Symptom Progression 6 month follow-up | 6 months post baseline
  Survey asking about disease diagnosis, testing, treatments, and symptom progression
IPF Symptom Progression 9 month follow-up | 9 months post baseline
  Survey asking about disease diagnosis, testing, treatments, and symptom progression

CONTACTS AND LOCATIONS:
Overall Officials: Suyash Shringarpure, Principal Investigator — 23andMe, Inc.
Locations (1):
- 23andMe, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided